CLINICAL TRIAL: NCT05152472
Title: A Prospective, Randomized, Multicenter, Comparative Study of the Efficacy of Imatinib Resumption Combined With Atezolizumab Versus Imatinib Resumption Alone in Patients With Unresectable Advanced Gastrointestinal Stromal Tumors (GIST) After Failure of Standard Treatments
Acronym: ATEZOGIST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET19-075- ATEZOGIST
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-02

CONDITIONS: Unresectable Gastrointestinal Stromal Tumor (GIST); Locally Advanced Gastrointestinal Stromal Tumor (GIST); Metastatic Gastrointestinal Stromal Tumor
Keywords: Oncology; Imatinib; Atezolizumab; Immunotherapy; Phase II; Unresectable Gastrointestinal Stromal Tumor; Locally Advanced Gastrointestinal Stromal Tumor; Metastatic Gastrointestinal Stromal Tumor; GIST; Tyrosine kinase inhibitor; Progression-Free Survival; Best Response Rate; Objective Response Rate; Time to Treatment Failure; Overall Survival; Quality of Life; Tolerability; Randomization
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasms | interventions — atezolizumab; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imatinib + Atezolizumab (Experimental): Imatinib per os 400 mg daily continuously associated with intravenous administrations of atezolizumab at the fixed dose of 1 200 mg every 3 weeks (up to 12 months)
  Interventions: Drug: Atezolizumab 1200 mg; Drug: Imatinib 400 MG
- Imatinib alone (Active Comparator): Imatinib alone, per os 400 mg daily continuously (up to 12 months)
  Interventions: Drug: Imatinib 400 MG

INTERVENTIONS:
Drug: Atezolizumab 1200 mg — (Intravenous administration)
  Other Names: Tecentriq®
  Arms: Imatinib + Atezolizumab
Drug: Imatinib 400 MG — (Per os)
  Other Names: Glivec®

SUMMARY:
This trial is a prospective, randomized (1:1 ratio), multicenter, comparative and phase II study, conducted in patients with unresectable advanced gastrointestinal stromal tumors (GIST) after failure of imatinib (disease progression),sunitinib and regorafenib (either disease progression or intolerance)

In the first arm, patients will be treated with imatinib + atezolizumab (experimental arm), whereas in the second arm, patients will be treated with imatinib alone (control arm).

The comparison between this two arms will allow to compare whether or not atezolizumab and imatinib is efficient for disease control, in terms of Progression-Free Survival improvement.

DETAILED DESCRIPTION:
This is a prospective, randomized (1:1 ratio), multicenter, comparative and phase II trial.

Patients with unresectable advanced gastrointestinal stromal tumors (GIST) will be accrued after the failure of standard treatments (imatinib, sunitinib and regorafenib) :

* For imatinib, failure is defined as disease progression
* For sunitinib and regorafenib, failure is defined as disease progression and/or intolerance

Randomization (1:1 ratio) will be stratified according to:

* The tumor KIT (exon 11) mutational status: wild type or mutated

STUDY TREATMENTS :

During the treatment period (12 months maximum), all patients will receive either:

* Imatinib per os 400 mg daily continuously associated with intravenous administrations of atezolizumab at the fixed dose of 1200 mg every 3 weeks (experimental arm)
* Or imatinib alone, per os 400 mg daily continuously (control arm)

The comparison between this two arms will allow to compare whether or not atezolizumab and imatinib is efficient for disease control, in terms of Progression-Free Survival improvement.

STATISTICAL ANALYSIS :

A total of 110 patients will be randomized (55 per arm).

It is expected a 6-month PFS rate of 10% in the standard arm (imatinib alone). Thus, a 6-month PFS-rate of 30% is a clinically significant target for patient treated with imatinib associated to immunotherapy.

An interim safety analysis is planned to be conducted after 6-month follow-up of the 12th patient has been randomized (approximately 6 patients by arm).

PFS will be estimated using the Kaplan-Meier method, and will be described in terms of median PFS along with the associated 2-sided 95% CIs for the estimates.

PFS distributions will be compared between the 2 study arms using a stratified Log-Rank test by tumor mutational status of KIT - exon 11 (stratification factors used for the randomisation).

A statistical interim analysis will be conducted after 50 events (PFS). Predefined stopping rules for futility will be applied to state on the continuation of the trial.

DATA ENTRY, DATA MANAGEMENT AND STUDY MONITORING :

All the data concerning the patients will be recorded in the electronic case report form (eCRF) throughout the study. Serious adverse event (SAE) and Adverse Event of Specific Interest (AESI) reporting will be also paper-based by e-mail and/or Fax.

The sponsor will perform the study monitoring and will help the investigators to conduct the study in compliance with the clinical trial protocol, Good Clinical Practices (GCP) and local law requirements.

ELIGIBILITY:
INCLUSION CRITERIA :

I1. Male or female ≥ 18 years at the day of consenting to the study;

I2. Patients must have histologically confirmed diagnosis of GIST (within the French Reference Network in Pathology of Sarcomas - RRePS network); Nota Bene: mutational status and level of expression of PD1/PD-L1 will not be considered as selection criteria but will be studied as endpoints for translational objectives.

I3. Locally advanced or metastatic disease confirmed as measurable according to the RECIST V1.1 (Appendix 1);

I4. Patients who previously failed to at least imatinib, sunitinib and then regorafenib. Failure is defined for Imatinib as progressive disease, and for sunitinib and regorafenib as progressive disease and/or intolerance;

I5. Performance Status of the ECOG of 0 or 1;

I6. Adequate bone marrow and organ function defined by the following laboratory results:

a. Bone marrow: i. Hemoglobin ≥ 9.0 g/dl, ii. Absolute Neutrophils Count (ANC) ≥ 1.5 G/l, iii. Lymphocytes count ≥ 0.5 G/l, iv. Platelets ≥ 100 G/l;

b. Coagulation: i. Prothrombin time ≤ 1.5 x Upper Limit of the Normal (ULN) for patients without therapeutic anticoagulation.

Patients with therapeutic anticoagulation must have stable dose of treatment.

c. Hepatic function: i. Total serum bilirubin ≤ 1.5 x ULN (except patients with Gilbert's syndrome who must have total serum bilirubin ≤ 3.0 x ULN), ii. Transaminases (ASAT/ALAT) ≤ 2.5 x ULN (or ≤ 5.0 x ULN in case of documented liver metastases) iii. Alkaline Phosphatases ≤ 2.5 x ULN (or ≤ 5.0 x ULN in case of documented bone metastases),

d. Renal function: i. Serum creatinine ≤ 1.5 x ULN or Cr. Cl. ≥ 40ml/min/1.73m² (MDRD or CKD-EPI formula);

I7. Willingness and ability to comply with the study requirements;

I8. Signed and dated informed consent indicating that the patient has been informed of all the aspects of the trial prior to enrolment;

I9. Women of childbearing potential are required to have a negative serum pregnancy test within 72 hours prior to study treatment start. A positive urine test must be confirmed by a serum pregnancy test;

I10. Women of childbearing potential and male patients must agree to use adequate highly effective contraception for the duration of study participation (Appendix 3);

I11. Patient must be covered by a medical insurance;

EXCLUSION CRITERIA :

E1. Prior malignancy within the last 3 years except for locally curable disease with no sign of relapse;

E2. Patients in whom imatinib had been already reintroduced after sunitinib as second line;

E3. Known D842V mutation in Exon 18 of PDGFRA;

E4. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-cytotoxic T lymphocyte-associated protein 4 , anti-TIGIT, anti PD-1,and anti PD-L1 therapeutic antibodies;

E5. Any approved anticancer therapy (chemotherapy, hormonal therapy or radiotherapy) or treatment with any investigational product within 2 weeks or within 5 elimination half-lives (whichever is longer) prior to study treatments start;

E6. Residual adverse events from prior anticancer therapy that has not resolved to grade ≤1, except for alopecia and lab values (provided that inclusion criteria described in section 6.1 are met);

E7. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.

Asymptomatic patients with treated CNS lesions are eligible, provided that all of the following criteria are met:

* Measurable disease, per RECIST v1.1, must be present outside the CNS.
* The patient has no history of intracranial hemorrhage or spinal cord hemorrhage.
* The patient has not undergone stereotactic radiotherapy within 7 days prior to randomization, whole-brain radiotherapy within 14 days prior to randomization, or neurosurgical resection within 28 days prior to randomization.
* The patient has no ongoing requirement for corticosteroids as therapy for CNS disease. Anticonvulsant therapy at a stable dose is permitted.
* Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord).
* There is no evidence of interim progression between completion of CNS-directed therapy and randomization.
* Spinal cord compression not definitively treated with surgery and/or radiation, and/or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for 2 weeks prior to screening.
* History of leptomeningeal disease.

E8. Patients using or require to use while on the study of any prohibited concomitant and/or concurrent medications (see section "Prohibited concomitant/concurrent treatments) :

* Live, attenuated vaccines within 28 days prior to enrolment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines, and are not allowed during the study active period.
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to C1D1, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:
* Patients who receive acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor confirmation.
* Patients who receive mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroid.
* Systemic immunostimulatory agents (including, but not limited to, interferons and IL-2) are prohibited within 4 weeks or five half-lives of the drug (whichever is longer) prior to C1D1.
* Traditional herbal medicines since the ingredients of many herbal medicines are not fully studied and their use may result in unanticipated drug-drug interactions that may cause or confound assessment of toxicity,

E9. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix 4 for a more comprehensive list of pre-existing autoimmune diseases and immune deficiencies), with the following exceptions:

* Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
* Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
* Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
* Rash must cover less than 10% of body surface area
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months

E10. History of severe allergic / anaphylactic reaction or other hypersensitivity reactions to:

* chimeric or humanized antibodies or fusion proteins,
* biopharmaceuticals produced in Chinese hamster ovary cells, any active substance or to any of the chemical excipients of atezolizumab (refer to its IB) or imatinib (refer to its respective SmPC)

E11. Patients with active infectious disease:

* severe infections within 4 weeks prior to randomisation including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia,
* active infection requiring or have required treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection) are eligible for the study.
* active B or C hepatitis infection, Note: Patients with past Hepatitis B Virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for Hepatitis C Virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* active tuberculosis
* HIV infection

E12. Active or prior history of primary immunodeficiency;

E13. Major surgical procedure within 28 days prior to study treatments start, or need for a major surgery during the course of the study;

E14. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within :

* 6 months after the final dose of study treatment for patients included in the standard arm (imatinib alone)
* 11 months after the final dose of study treatment for patients included in the experimental arm (imatinib + atezolizumab) Women of childbearing potential must have a negative pregnancy test result within 72 hours prior to treatment start (any urine positive pregnancy test must be confirmed by a serum pregnancy test prior to treatment start);

E15. Patient that impairs their ability to swallow and retain imatinib or with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of imatinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)

E16. Clinically significant unrelated systemic illness (e.g., significant cardiac, pulmonary, hepatic, or other organ dysfunction) that would compromise the patient's ability to tolerate study treatment or would likely interfere with study procedures or results.

E17. Patients under tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 48 months
  Time from the date of randomization to the date of first disease progression, or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Best Response Rate (BRR) | 48 months
  The best response from randomization : Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD)
Objective Response Rate (ORR) | 48 months
  The proportion of patients with a best overall response of CR or PR during the study
Time to Treatment Failure (TTF) | 48 months
  The time from the date of randomization to the date of permanent study treatments discontinuation (any cause, including death, progression, discontinuation of treatment due to progression, toxicity or start of a new anticancer therapy and withdrawal of consent)
Overall Survival (OS) | 48 months
  The time from the date of randomization to the date of death due to any cause
Quality of Life (QoL) | Up to 12 months
  Assessed using the EORTC QLQ-C30 questionnaire
Tolerability profile | 48 months
  Described through the incidence and severity of drug-related AEs (AE, SAE, SUSAR, new safety issue) according to the National Cancer Institute Common Terminology Criteria for Adverse Event Version 5 (NCI-CTC AE V5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi BRAHMI, MD, Principal Investigator — Centre Leon Berard
Locations (13):
- France (13):
  - Centre Léon Bérard, Lyon, Rhône
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Hôpital de La Timone, Marseille
  - Centre Antoine Lacassagne, Nice
  - CHU Poitiers, Poitiers
  - Hôpital Robert Debré, Reims
  - Centre Eugène Marquis, Rennes
  - Institut de cancérologie de l'Ouest, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - ICANS CHRU de Strasbourg, Strasbourg
  - Chru Tours, Tours
  - Institut Gustave Roussy, Villejuif